CLINICAL TRIAL: NCT03164785
Title: Efficacy and Safety of Jinshuibao Capsule as Add-on Therapy to Angiotensin II Receptor Blockers on Diabetic Kidney Disease in Patients With Type 2 Diabetes Mellitus
Brief Title: Efficacy and Safety of Jinshuibao Capsule on Diabetic Kidney Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Zhiguang Zhou, Head of Endocrinology Department, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JSB201601
Record Dates: First submitted 2017-05-08; First posted 2017-05-24 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Type 2 Diabetes Mellitus; Diabetic Kidney Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies | interventions — CME-1 polysaccharide, Cordyceps sinensis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Experimental): Treatment：subjects receive Jinshuibao Capsule. ARB will be continued as a routine therapy.
  Counseling: subjects will follow through regular check-up and receive lifestyle and other diabetes treatment counseling
  Interventions: Drug: Jinshuibao Capsule
- Control Group (No Intervention): Patients receive a standard dose of ARB drug as a routine therapy. Counseling: subjects will follow through regular check-up and receive lifestyle and other diabetes treatment counseling

INTERVENTIONS:
Drug: Jinshuibao Capsule — 1.98g t.i.d. p.o. for 6 months
  Other Names: Jinshuibao Jiaonang; Cordyceps sinensis; Artificial Cordyceps sinensis powder
  Arms: Treatment Group

SUMMARY:
The purpose of this study is to investigate the therapeutic effect and safety of Jinshuibao Capsule on diabetic kidney disease in T2DM patients.

DETAILED DESCRIPTION:
Diabetic Kidney Disease (DKD) is one of the most important microvascular complications of diabetes and is the leading cause of end-stage renal disease. Intensive glycemic and blood pressure control, combined with renin - angiotensin system blocking therapy (including ACEI and ARB drugs), has to a certain extent, delayed the progression of DKD, but still cannot completely block its development. Cordyceps sinensis is a traditional Chinese medicine and Jinshuibao Capsule is its artificial preparation, with the effect of renoprotection. However, its clinical application in diabetic kidney disease is not well-defined so far. The aim of this study is to investigate the potential use of Jinshuibao Capsule on microalbuminuria in T2DM.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with written informed consent.
2. Type 2 diabetes according to 1999 WHO criteria.
3. Age: 30-75 years.
4. HbA1c < 11%.
5. Stage III diabetic kidney disease:

   5.1 microalbuminuria: 30 mg / g < urinary albumin creatinine ratio (ACR) < 300 mg / g, positive for at least two in three times.

   5.2 renal function: eGFR ≧ 30 ml / min / 1.73 ㎡.
6. Stable use of a standard dose of angiotensin II receptor blocker ≧ 3 months.
7. Childbearing-age women with contraceptive measures.

Exclusion Criteria：

1. Type 1 Diabetes Mellitus.
2. Non-diabetic urinary system diseases (Urinary tract obstruction, bladder emptying disorders, severe benign prostatic hyperplasia, renal vascular disease, post-renal transplantation, active urinary tract infection,etc.)
3. Other serious diseases [severe hypertension ((defined as SBP > 200 mmHg and/or DBP > 110 mmHg, or requiring ≧3 anti-hypertensive drugs simultaneously), cardiovascular and cerebrovascular events within 6 months, autoimmune diseases implicating the urinary system, chronic or acute pancreatitis, malignancy, hepatic abnormalities (transaminase ≧ 3.0 x UNL), severe gastrointestinal diseases, other endocrine diseases affecting the urinary system, etc.]
4. Allergic to Cordyceps sinensis, use of ACEIs, any use of Cordyceps sinensis preparations, systemic glucocorticoid treatment ≧ 7 days within a month, use of nephrotoxic drugs within 3 months, alcohol or psychotropic drug dependence, etc.
5. Presence of acute metabolic disorders (DKA,HHS); history of surgery, severe trauma and other stress conditions.
6. Female patients who are pregnant or breastfeeding. Any medical condition that, in the opinion of the investigator, will interfere with participation in the trial.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2020-09-26 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Change in urine albumin creatine ratio (ACR). | Baseline and 1,2,3,6 months.
  First morning urine (10-15ml) of the subject is collected with a clean urine collection tube (or vial).

SECONDARY OUTCOMES:
The incidence of ≧30% decline in eGFR from baseline. | half a year
  Monitoring changes in glomerular functions measured in estimated glomerular filtration rate (eGFR) [CKD-EPI creatinine-cystatin equation (2012)].
Change in urine α1-microglobulin. | Baseline and 1,2,3,6 months.
Change in urine β2-microglobulin. | Baseline and 1,2,3,6 months.
Change in urine N-acetyl-β-D-glucosidase. | Baseline and 1,2,3,6 months.
Change in urine neutrophil gelatinase-associated lipocalin. | Baseline and 1,2,3,6 months.
Change in inflammation level. | Baseline and 1,2,3,6 months.
  Change in hs-CRP level.
Change in HbA1c. | Baseline and 1,3,6 months.
Change in blood pressure control. | Baseline and 1,2,3,6 months.
Change in blood lipids. | Baseline and 1,3,6 months.
Life quality evaluation | Baseline and 6 months.
  Change in SF-36 Scale score.
Incidence of Treatment-Emergent Adverse Events | half a year
  Treatment-related adverse events as assessed by deterioration of liver functions with other reasons excluded, self-report of gastrointestinal symptoms associated with drug intake, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiguang Zhou, MD/PhD, Principal Investigator — Second Xiangya Hospital of Central South University
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No
The results belongs to the principal investigator and collaborators.